CLINICAL TRIAL: NCT04354948
Title: The Influence of Pain on Exercise-Induced Hypoalgesia in Healthy Subjects: A Randomized Controlled Trial
Brief Title: Influence of Pain on Exercise-induced Hypoalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Henrik Bjarke Vægter, Associate Professor in Physiotherapy, Odense University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S-20190081
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Pain
Keywords: Exercise-induced hypoalgesia; Pressure pain threshold; hypertonic saline
MeSH Terms: conditions — Pain | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: This study is a 2-arm randomized controlled cross-over trial with 1 week between arms
Who Masked: Investigator
Masking Description: The researcher responsible for the statistical analyses are blinded to arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain (hypertonic saline) (Experimental): Injection (1 ml) of painful hypertonic saline (5.8%) prior to performance of the 3 min wall squat exercise
  Interventions: Behavioral: Pain (hypertonic saline)
- No pain (Hypotonic saline) (Placebo Comparator): Injection (1 ml) of non-painful isotonic saline (0.9%) prior to performance of the 3 min wall squat exercise
  Interventions: Behavioral: No pain (Hypotonic saline)

INTERVENTIONS:
Behavioral: Pain (hypertonic saline) — A bolus injection (1 ml) of hypertonic saline (5.8%) is injected into the right quadriceps femoris of the quadriceps femoris muscle 1 minute before performance of the 3 min wall squat exercise
  Arms: Pain (hypertonic saline)
Behavioral: No pain (Hypotonic saline) — A bolus injection (1 ml) of isotonic saline (0.9%) is injected into the right quadriceps femoris of the quadriceps femoris muscle 1 minute before performance of the 3 min wall squat exercise
  Arms: No pain (Hypotonic saline)

SUMMARY:
The purpose of this study is to investigate how acute pain induced by hypertonic saline prior to exercise influence the magnitude of exercise-induced hypoalgesia after a 3 min isometric wallsquat exercise in healthy subjects. The study is a single blinded (investigator) randomized cross-over trial The results from the study may be of great importance to the understanding of exercise-induced hypoalgesia, and whether the presence of pain affects the effects of exercise.

DETAILED DESCRIPTION:
Exercise is recommended to promote and maintain health and as treatment for more than 25 chronic diseases and pain conditions.

The mechanisms underlying pain relief of exercise are largely unknown but may be related to the modulation of central descending pain inhibitory pathways after acute exercise bouts. Exercise-induced hypoalgesia (EIH) is typically assessed as the temporary change in PPTs after a short acute exercise bout and EIH is seen as a proxy of descending pain inhibitory control. In general, EIH seems hypoalgesic (functional) in asymptomatic subjects. A hyperalgesic (impaired) EIH response has been reported in different chronic pain populations, although a functional EIH response also has been reported in subgroups of knee osteoarthritis patients. This implies differences in the acute response to exercise between healthy (pain-free) subjects and chronic pain patients, but it is still unknown whether the presence of pain itself affects the pain alleviating response (i.e. the EIH response) to acute exercise.

It is hypothesized that acute pain will decrease the EIH response magnitude following hypertonic saline injection compared with the control injection. This study will increase the insight into the EIH mechanisms in healthy subjects in general, and how the presence of pain affects the body's own ability to modulate pain during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Pain-free
* Understands and writes Danish

Exclusion Criteria:

* Pregnancy
* Previous addictive behavior defined as abuse of hash, opioids or other euphoric substances.
* Previous painful or mental illnesses, neurological or circulatory diseases in the form of heart or lung disease.
* Surgery within last 3 months
* Pain on the days of testing
* Pain for more than 2 weeks within the last 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold at the right quadriceps muscle where injection is performed. | Before and after the 3 minutes wall squat
  Between group comparison of the primary outcome, which is change in pressure pain threshold at the right quadriceps muscle from before wall squat to after wall squat. Pressure pain threshold is measured with a hand held pressure algometer.

SECONDARY OUTCOMES:
Pressure pain threshold at the non-dominant trapezius muscle | Before and after the 3 minutes wall squat
  Between group comparison of the secondary outcome, which is change in pressure pain threshold at the left trapezius muscle from before wall squat to after wall squat. Pressure pain threshold is measured with a hand held pressure algometer.
Pressure pain threshold at the left quadriceps muscle where injection is not performed. | Before and after the 3 minutes wall squat
  Between group comparison of the secondary outcome, which is change in pressure pain threshold at the left quadriceps muscle from before wall squat to after wall squat. Pressure pain threshold is measured with a hand held pressure algometer.
Pain Intensity in thighs | Assessed before and immediately after hypertonic and isotonic saline injection as well as after 1, 2 and 3 min of wall squat, and immediately after the end of wall squat
  Pain intensity in both thighs are assessed with numerical rating scales with 0 = no pain and 10 = maximal pain.

OTHER OUTCOMES:
Pressure pain threshold | At baseline on both days before saline injections
  Cuff pressure pain threshold (cPPT) is assessed using a computer-controlled cuff pressure algometer (CPAR, NociTech, Denmark,). A 13-cm wide silicone tourniquet cuff is wrapped around the right lower leg with an 8-cm distance to the tibial tuberosity. The cuff pressure is increased with a rate of 1 kPa/s and the maximal pressure limit is 100 kPa. The participants use an electronic visual analog scale (VAS) to rate the pressure-induced pain intensity and a button to release the pressure. Zero- and 10-cm extremes on the VAS were defined as "no pain" and as "maximal pain," respectively. The participants are instructed to rate the pain intensity continuously on the electronic VAS from when the pressure was defined as first sensation of pain and to press the pressure release button when the pain was intolerable. The pressure value when the subject rated the sensation of pain as 1 cm on the VAS was defined as the cPPT.
Pressure pain tolerance | At baseline on both days before saline injections
  Cuff pressure pain tolerance (cPTT) is assessed using a computer-controlled cuff pressure algometer (CPAR, NociTech, Denmark,). A 13-cm wide silicone tourniquet cuff is wrapped around the right lower leg with an 8-cm distance to the tibial tuberosity. The cuff pressure is increased with a rate of 1 kPa/s and the maximal pressure limit is 100 kPa. The participants use an electronic visual analog scale (VAS) to rate the pressure-induced pain intensity and a button to release the pressure. Zero- and 10-cm extremes on the VAS were defined as "no pain" and as "maximal pain," respectively. The participants are instructed to rate the pain intensity continuously on the electronic VAS from when the pressure was defined as first sensation of pain and to press the pressure release button when the pain was intolerable. The pressure value when the subject terminates the pressure inflation is defined as the cPTT.
Temporal summation of pain | At baseline on both days before saline injections
  Temporal summation of pain (TSP) is assessed at the right lower leg with computer-controlled cuff algometry. Ten repeated cuff pressure stimulations lasting 1 second each (1 sec breaks in between) are induced to assess TSP. Stimulations are delivered by rapid inflation of the cuff with an intensity equivalent to the pressure pain tolerance. Subjects rate the pain intensity on an electronic VAS continuously during the sequential stimulation without returning the VAS to zero between stimulations. VAS scores immediately after each stimulus are extracted, and TSP is calculated as the ratio of the last 3 stimulations to the first four stimulations, with positive values indicating an increase in pain intensity ratings during the repeated stimulation.
International Physical Activity Questionnaire (IPAQ) | Baseline of first session
  The IPAQ is suitable for adults between 15 and 69 years of age and is used for sample surveillance of physical activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik B Vægter, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Pain Center, University Hospital Odense, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen S, Petersen KK, Sloth E, Manum LA, McDonald AK, Andersen PG, Vaegter HB. Hypoalgesia after exercises with painful vs. non-painful muscles in healthy subjects - a randomized cross-over study. Scand J Pain. 2021 Dec 27;22(3):614-621. doi: 10.1515/sjpain-2021-0161. Print 2022 Jul 26. PMID 34958721